CLINICAL TRIAL: NCT03629054
Title: Bioequivalence of a Low Strength Fixed Dose Combination Tablet of Empagliflozin/Linagliptin/Metformin Extended Release Compared to the Free Combination of Empagliflozin, Linagliptin, and Metformin Extended Release Tablets Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: This Study in Healthy People Tests Whether Taking a Low Strength of Empagliflozin, Linagliptin, and Metformin Together in 1 Pill is the Same as Taking Them in Separate Pills
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1361-0011; 2018-001266-42 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test treatment (T) (Experimental): Low strength empagliflozin/linagliptin/metformin XR fixed dose combination tablet
  Interventions: Drug: Empagliflozin, Metformin HCl, Linagliptin (fixed dose combination)
- Reference treatment (R) (Experimental): Single tablets of empagliflozin + linagliptin + metformin XR
  Interventions: Drug: Empagliflozin; Drug: Linagliptin; Drug: Metformin HCl

INTERVENTIONS:
Drug: Empagliflozin, Metformin HCl, Linagliptin (fixed dose combination) — single dose
  Other Names: TRIJARDY® XR
  Arms: Test treatment (T)
Drug: Empagliflozin — single dose
  Arms: Reference treatment (R)
Drug: Linagliptin — single dose
  Arms: Reference treatment (R)
Drug: Metformin HCl — single dose
  Arms: Reference treatment (R)

SUMMARY:
The primary objective of this trial is to establish the bioequivalence of two empagliflozin/linagliptin/metformin extended release (XR) fixed dose combination (FDC) tablets (Test, T) compared with the same doses of the individual components given in separate tablets (Reference, R) when administered together after a high-fat, high-calorie meal.

The assessment of safety and tolerability will be the secondary objective of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Female subjects of childbearing potential willing to use adequate contraception.
* Further inclusion criteria apply

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to include healthy participants in this randomised, open-label, two-way crossover trial with 2 treatments (test treatment (T) and reference treatment (R)) and 2 treatment sequences (TR or RT) in order to compare the treatment T to the treatment R under fed conditions. They were recruited from the volunteers' pool of the study site.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial and to ensure that all participants met all inclusion/exclusion criteria. Participants were not to be included in the trial if any of the specific exclusion criteria were met.
Groups:
- Test Treatment (T)/ Reference Treatment (R): Participants were administered 2 fixed dose combination (FDC) coated tablets of 5 milligram (mg) empagliflozin/ 2.5 mg linagliptin/ 1000 mg metformin extended release (XR) orally as a single dose in the fed state in period 1, followed by the free combination of 1 film-coated tablet of 10 mg empagliflozin, 1 film-coated tablet of 5 mg linagliptin and 4 film-coated tablets of 500 mg metformin XR orally as single dose in the fed state in period 2. The T and R treatments were separated by a washout period of at least 35 days.
- Reference Treatment (R)/ Test Treatment (T): Participants were administered the free combination of 1 film-coated tablet of 10 mg empagliflozin, 1 film-coated tablet of 5 mg linagliptin and 4 film-coated tablets of 500 mg metformin XR orally as single dose in the fed state in period 1 and followed by 2 FDC coated tablets of 5 mg empagliflozin/ 2.5 mg linagliptin/ 1000 mg metformin XR orally as a single dose in the fed state in period 2. The T and R treatments were separated by a washout period of at least 35 days.
Period: Period 1 (4 Days)
Arm/Group | Test Treatment (T)/ Reference Treatment (R) | Reference Treatment (R)/ Test Treatment (T)
Started (Started are treated) | 15 (Started this period) | 15 (Started this period)
Completed | 15 | 15
Not Completed | 0 | 0
Period: Wasout Period (35 Days)
Arm/Group | Test Treatment (T)/ Reference Treatment (R) | Reference Treatment (R)/ Test Treatment (T)
Started (Started are treated) | 15 (Started this period) | 15 (Started this period)
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2 (4 Days)
Arm/Group | Test Treatment (T)/ Reference Treatment (R) | Reference Treatment (R)/ Test Treatment (T)
Started | 15 (Started this period) | 15 (Started this period)
Treated | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS): TS included all subjects who were documented to have received at least one dose of study drug.
Groups:
- Test Treatment (T)/ Reference Treatment (R): Participants were administered 2 fixed dose combination (FDC) coated tablet of 5 milligram(mg) empagliflozin/ 2.5 mg linagliptin/ 1000 mg metformin extended release (XR) orally in the fed state in period 1, followed by free combination of 1 film-coated tablet of 10 mg empagliflozin, 1 film-coated tablet of 5 mg linagliptin and 4 film-coated tablets of 500 mg metformin XR in the fed state in period 2. The T and R treatments were separated by a washout period of at least 35 days.
- Total: Total of all reporting groups
Arm/Group | Test Treatment (T)/ Reference Treatment (R) | Reference Treatment (R)/ Test Treatment (T) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (7.6) | 41.5 (9.7) | 44.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Empagliflozin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, Area under the concentration-time curve of the empagliflozin in plasma over the time interval from 0 to the last quantifiable data point is presented. Standard error (SE) is a geometric SE.
Time Frame: Pharmacokinetic (PK) samples were collected 1:30 hours:minutes (h:m) pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 10:00, 12:00, 24:00, 34:00, 48:00 and 72:00 h:m after drug administration.
Population: Pharmacokinetic parameter set (PKS): PKS included all subjects in the treated set (TS) who provided at least one primary or secondary PK parameter that was not excluded due to protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: nanomole*hour/litre (nmol*h/L)
Groups:
- Test Treatment (T): Participants were administered 2 FDC coated tablets of 5 mg empagliflozin/ 2.5 mg linagliptin/ 1000 mg metformin XR orally as a single dose in the fed state.
- Reference Treatment (R): Participants were administered the free combination of 1 film-coated tablet of 10 mg empagliflozin, 1 film-coated tablet of 5 mg linagliptin and 4 film-coated tablets of 500 mg metformin XR orally as single dose in the fed state.
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nanomole*hour/litre (nmol*h/L) | 2134.53 (1.03) | 2125.57 (1.03)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); An ANOVA model on the logarithmic scale including fixed effects for 'sequence', 'period' and 'treatment' and random effect for 'subject within sequence'; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (gMean) (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 100.42, 90% CI 2-sided [98.17 to 102.72], Standard Error of Mean 4.8 — gMean ratio = T/R. Standard error of the mean is actually intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Area Under the Concentration-time Curve of the Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, Area under the concentration-time curve of the metformin in plasma over the time interval from 0 to the last quantifiable data point is presented. Standard error (SE) is a geometric SE.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanogram*h/mL (ng*h/mL)
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nanogram*h/mL (ng*h/mL) | 21687.12 (1.04) | 22748.21 (1.04)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 95.34, 90% CI 2-sided [91.58 to 99.24], Standard Error of Mean 8.5 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

3. Primary Outcome: Area Under the Concentration-time Curve of the Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours (h) (AUC0-72)
Description: AUC0-72, area under the concentration-time curve of the linagliptin in plasma over the time interval from 0 to 72 h is presented. SE is a geometric SE.
Time Frame: PK samples were collected 1:30 h:m pre-dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 10:00, 12:00, 24:00, 34:00, 48:00 and 72:00 h:m after drug administration.
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nmol*h/L | 270.19 (1.03) | 269.77 (1.03)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 100.16, 90% CI 2-sided [96.17 to 104.31], Standard Error of Mean 8.6 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

4. Primary Outcome: Maximum Measured Concentration of the Empagliflozin in Plasma (Cmax)
Description: Cmax, maximum measured concentration of the empagliflozin in plasma is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanomole/Litre (nmol/ L)
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nanomole/Litre (nmol/ L) | 209.67 (1.05) | 226.50 (1.05)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p = 0.0029, ANOVA; Adjusted gMean ratio = 92.57, 90% CI 2-sided [85.21 to 100.57], Standard Error of Mean 17.9 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

5. Primary Outcome: Maximum Measured Concentration of the Linagliptin in Plasma (Cmax)
Description: Cmax, maximum measured concentration of the linagliptin in plasma is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanomole/Litre (nmol/ L)
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nanomole/Litre (nmol/ L) | 7.02 (1.05) | 7.21 (1.05)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p = 0.0001, ANOVA; Adjusted gMean ratio = 97.33, 90% CI 2-sided [89.99 to 105.26], Standard Error of Mean 16.9 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

6. Primary Outcome: Maximum Measured Concentration of the Metformin in Plasma (Cmax)
Description: Cmax, maximum measured concentration of the metformin in plasma is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanogram/ millilitre (ng/ mL)
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nanogram/ millilitre (ng/ mL) | 1853.03 (1.04) | 1767.69 (1.04)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 104.83, 90% CI 2-sided [98.56 to 111.50], Standard Error of Mean 13.2 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

7. Secondary Outcome: Area Under the Concentration-time Curve of the Empagliflozin Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of the empagliflozin in plasma over the time interval from 0 extrapolated to infinity is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nmol*h/L | 2182.26 (1.03) | 2166.54 (1.03)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 100.73, 90% CI 2-sided [98.33 to 103.18], Standard Error of Mean 5.1 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

8. Secondary Outcome: Area Under the Concentration-time Curve of the Linagliptinin Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of the linagliptin in plasma over the time interval from 0 extrapolated to infinity is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
nmol*h/L | 471.40 (1.05) | 455.13 (1.05)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 103.57, 90% CI 2-sided [96.90 to 110.71], Standard Error of Mean 14.3 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

9. Secondary Outcome: Area Under the Concentration-time Curve of the Metformin Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of the metformin in plasma over the time interval from 0 extrapolated to infinity is presented. SE is a geometric SE.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Standard Error); unit: ng*h/mL
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
ng*h/mL | 22288.72 (1.04) | 23280.48 (1.04)
Statistical Analysis 1: Comparison: Test Treatment (T) vs Reference Treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The assessment of bioequivalence was based upon two-sided 90% CIs for the ratios of the geometric means (T/R); p < 0.0001, ANOVA; Adjusted gMean ratio = 95.74, 90% CI 2-sided [92.29 to 99.32], Standard Error of Mean 7.8 — gMean ratio = T/R. Standard Error of the mean is actually intra-individual gCV

10. Secondary Outcome: Percentage of Patients With Drug-related Adverse Events (AEs)
Description: Percentage of patients with investigator defined drug-related AEs are presented.
Time Frame: All adverse events (AEs) which occurred through the treatment phase and throughout the residual effect period (REP), up to 7 days.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Test Treatment (T) | Reference Treatment (R)
Number analyzed (Participants) | 29 | 30
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) which occurred through the treatment phase and throughout the residual effect period (REP), up to 7 days. All cause mortality and serious AEs are considering the entire duration of the trial, 49 days.
Arm/Group | Test Treatment (T) | Reference Treatment (R)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 8/29 | 6/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Treatment (T) (N=29) | Reference Treatment (R) (N=30)
Nausea (Gastrointestinal disorders) | 4 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT03629054/SAP_000.pdf
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03629054/Prot_001.pdf